CLINICAL TRIAL: NCT00638677
Title: Bifidobacterium Lactis BB12 and Xylitol Delivered With a Novel Slow-release Pacifier
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Chr Hansen A/S (Unknown); Fennobon oy, Karkkila, Finland (provides the tablets for the pacifier) (Unknown); Plastone Oy, Konnevesi, Finland (provides the pacifiers) (Unknown)
Responsible Party: Principal Investigator, Eva Soderling, Associate professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pacifierstudy20/8/2003; No ISRCTN or NIH grants
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Dental Caries; Infectious Diseases
Keywords: Oral microbiology
MeSH Terms: conditions — Dental Caries; Communicable Diseases | interventions — Sorbitol; Xylitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Sorbitol tablet
  Interventions: Dietary Supplement: Sorbitol
- 2 (Placebo Comparator): Xylitol tablet
  Interventions: Dietary Supplement: Xylitol
- 3 (Active Comparator): Xylitol + BB12 tablet
  Interventions: Dietary Supplement: Xylitol + BB12

INTERVENTIONS:
Dietary Supplement: Sorbitol — Sorbitol tablet delivered with a slow-release pacifier starting 1 mo after delivery and lasting max 2 years
  Other Names: Xylitol; Bifidobacterium lactis
  Arms: 1
Dietary Supplement: Xylitol + BB12 — Xylitol + BB12 tablet delivered with a slow-release pacifier starting 1 mo after delivery and continuing max 2 years
  Other Names: Sorbitol; Bifidobacterium lactis
  Arms: 3
Dietary Supplement: Xylitol — Xylitol+BB 12 delivery with a pacifier max until 2 years
  Other Names: Sorbitol; Bifidobacterium lactis
  Arms: 2

SUMMARY:
Aims:

1. To develop a food supplement containing a health-promoting probiotic bacteria (B. lactis BB12) and xylitol to be administered with a novel soft, possibly occlusion-friendly pacifier.
2. Test in a clinical study how feasible the method is and to study how the intervention affects caries occurrence.

Main hypothesis:

The administration of B. lactis BB12 and xylitol affects beneficially the dental health of the child.

DETAILED DESCRIPTION:
Xylitol is known to reduce counts of mutans streptococci (ms) as well as mother-child transmission of ms. Possibly xylitol delivered to infants could positively influence colonization/metabolism of ms. By combining in a food supplement xylitol and B. lactis BB12 (a well known probiotic bacteria) we may be able to positively affect both gut and oral colonization, reflected in both dental and general health (solid data available on the latter aim). Though B. lactis is in wide use in baby formulas and in in vitro tests it apparently is safe for the teeth, no clinical studies have looked at effects of its administration to infants on oral health. Our study aims to look at caries occurrence in infants who have received the xylitol + BB12 food supplement with a pacifier.

Recruiting of subjects to the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* The infant is healthy
* The family agrees to use the novel slow-release pacifier
* The infant starts to use the pacifier before the age of 3 months

Exclusion Criteria:

* The child is not healthy

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2004-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
MS colonization | 2 years

SECONDARY OUTCOMES:
Acute infectious diseases | 2 years
Caries occurrence | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Söderling, PhD, Principal Investigator — Assoc. Prof., University of Turku
Locations (1):
- Health Care Centre, Muurame and Korpilahti, Finland

REFERENCES:
- [Derived] Taipale T, Pienihakkinen K, Alanen P, Jokela J, Soderling E. Administration of Bifidobacterium animalis subsp. lactis BB-12 in early childhood: a post-trial effect on caries occurrence at four years of age. Caries Res. 2013;47(5):364-72. doi: 10.1159/000348424. Epub 2013 Apr 5. PMID 23571819